CLINICAL TRIAL: NCT07180043
Title: Clinical Predictors of Propranolol Responsiveness in Pediatric Migraine: A Prospective Observational Study
Brief Title: Propranolol for Pediatric Migraine: A Prospective Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri University (Other)
Responsible Party: Principal Investigator, Özge BAYKAN ÇOPUROĞLU, Asst. Prof., Kayseri University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KayseriUniversity; EC/IRB Number (Other: Tepecik Training and Research Hospital Ethics Committee)
Record Dates: First submitted 2025-09-04; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Migraine; Headache Disorders
Keywords: Pediatric Migraine; Propranolol; Behavioral Therapy
MeSH Terms: conditions — Headache Disorders | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Behavioral Therapy (Other): Participants received structured behavioral therapy including patient education, lifestyle guidance, and maintenance of a headache diary, without pharmacological prophylaxis.
  Interventions: Behavioral: Structured Behavioral Therapy
- Propranolol (Experimental): Participants received oral propranolol at 1-3 mg/kg/day in two divided doses for 12 weeks. Dose titration was performed based on clinical response and tolerance.
  Interventions: Drug: Propranolol

INTERVENTIONS:
Behavioral: Structured Behavioral Therapy — Structured patient education, lifestyle modification counseling, and headache diary maintenance without pharmacological prophylaxis.
  Arms: Structured Behavioral Therapy
Drug: Propranolol — Oral propranolol, 1-3 mg/kg/day in two divided doses, titrated according to response, for 12 weeks.
  Arms: Propranolol

SUMMARY:
This prospective, controlled clinical trial was conducted to evaluate the effectiveness of propranolol compared with structured behavioral therapy in pediatric patients diagnosed with primary migraine according to ICHD-3 criteria. A total of 178 children aged 6 to 16 years were enrolled between January 2021 and December 2023 at a tertiary pediatric neurology center.

Participants were allocated into two groups based on baseline Pediatric Migraine Disability Assessment (PedMIDAS) scores: Group 1 received standardized behavioral therapy, while Group 2 received propranolol at doses ranging from 1-3 mg/kg/day for 12 weeks. Primary outcomes included changes in PedMIDAS and Visual Analog Scale (VAS) scores. Secondary analyses investigated clinical and biochemical predictors of propranolol responsiveness, including benign paroxysmal vertigo, essential tremor, anxiety, vitamin D status, and vitamin B12 levels.

The study aims to provide evidence for a more personalized approach to migraine prophylaxis in children by integrating clinical, psychiatric, and nutritional predictors of treatment response.

DETAILED DESCRIPTION:
Migraine is among the most common neurological disorders in children and adolescents, often leading to significant disability, reduced school performance, and impaired quality of life. Although propranolol is frequently prescribed for pediatric migraine prophylaxis, previous studies have reported heterogeneous outcomes, and clinical predictors of treatment response remain unclear.

This prospective, controlled clinical trial was designed to assess the comparative effectiveness of propranolol and structured behavioral therapy in pediatric migraine patients and to identify predictors of response to propranolol. A total of 178 children, aged 6-16 years, diagnosed with primary migraine according to ICHD-3 criteria, were consecutively recruited at a tertiary pediatric neurology center between January 2021 and December 2023.

Participants were allocated into two groups based on baseline Pediatric Migraine Disability Assessment (PedMIDAS) scores:

Group 1 (n = 88) received structured behavioral therapy, including patient education, lifestyle guidance, and headache diary maintenance.

Group 2 (n = 90) received oral propranolol at doses of 1-3 mg/kg/day for 12 weeks, with adherence monitored through logs and follow-up calls.

The primary outcomes were changes in PedMIDAS and Visual Analog Scale (VAS) scores after 12 weeks. Secondary outcomes included identification of clinical, psychiatric, and biochemical predictors of treatment responsiveness. Particular attention was given to benign paroxysmal vertigo, essential tremor, anxiety traits, and micronutrient deficiencies (vitamin D and vitamin B12).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary migraine (with or without aura) according to ICHD-3 criteria
* Age between 6 and 16 years
* Minimum of 4 migraine attacks per month
* No history of prophylactic migraine therapy within the last 3 months
* Written informed consent obtained from parents or legal guardians

Exclusion Criteria:

* Secondary headaches due to underlying pathologies (e.g., tumors, infections, vascular malformations)
* Chronic systemic or psychiatric disorders (e.g., epilepsy, major depression)
* Contraindications to propranolol (e.g., asthma, cardiac conduction defects)
* Incomplete clinical data or loss to follow-up

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 178 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Pediatric Migraine Disability Assessment (PedMIDAS) Score | Baseline and Week 12
  Change in PedMIDAS score from baseline to 12 weeks, assessing migraine-related disability in pediatric patients. The PedMIDAS score ranges from 0 to 240, with higher scores indicating greater migraine-related disability. Lower scores reflect less disability and therefore a better outcome.
Change in Visual Analog Scale (VAS) Pain Score | Baseline and Week 12
  Change in VAS pain intensity score from baseline to 12 weeks, evaluating migraine pain severity. The VAS score ranges from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores represent worse pain severity, while lower scores indicate improvement.

SECONDARY OUTCOMES:
Responder Rate | Week 12
  Proportion of participants achieving ≥50% reduction in monthly migraine frequency compared with baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri University, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No